CLINICAL TRIAL: NCT07084220
Title: The Effect of Cognitive Tasks on Single Limb Balance
Status: Completed | Type: Observational
Sponsor: Towson University (Other)
Responsible Party: Principal Investigator, Lisa Custer, Associate Professor, Towson University
Other Study IDs: 1907054099
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2019-08

CONDITIONS: Chronic Ankle Instability, CAI; Healthy Participants
Keywords: dual-task; ankle; balance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control: * No previous history of ankle sprain on either limb
  * A score lower than 10 on the Identification of Functional Ankle Instability
  * Between 18-40 years old
  * Lower extremity injury-free for at least 3 months
  * No previous history of foot or ankle surgery on either limb
  * No known history of known foot or ankle fracture on either limb
  * No known neurological or vestibular disorders, or other medical conditions affecting balance, including ear infections
  * Does not have diabetes mellitus
  * No self-reported disability due to lower extremity pathology
- Chronic ankle instability: * Between 18-40 years old
  * Lower extremity injury-free for at least 3 months
  * No previous history of foot or ankle surgery on either limb
  * No known history of known foot or ankle fracture on either limb
  * No known neurological or vestibular disorders, or other medical conditions affecting balance, including ear infections
  * Does not have diabetes mellitus
  * No self-reported disability due to lower extremity pathology
  * A previous history of at least 1 lateral ankle sprain as reported on the Modified Ankle Instability Index
  * A score of 10 or higher on the Identification of Functional Ankle Instability

SUMMARY:
Purpose of the Study: The purpose of this study is to evaluate the effects of performing various cognitive tasks on balance in individuals with chronic ankle instability and healthy controls. Three different cognitive tasks will be performed while participants balance on one limb. Chronic ankle instability is defined as having a history of at least one ankle sprain and having residual effects. The specific aims of this study are to:

1. Determine if performing the cognitive tasks effect single limb balancing.
2. Determine which cognitive task, if any, has the greatest effect on single limb balance.

Participants will perform single-limb balancing with eyes open on the force plate while performing one of the four cognitive tasks. You will start with the control condition, the order of cognitive tasks will be random. Testing will occur on both limbs.

1. Each trial will last 1 minute. There will be at least a 30 second rest period between trials.
2. You will perform 3 trials of each cognitive task prior to moving on to the next task. There will be a 5 minute rest between cognitive tasks.
3. You will complete all testing on one limb (counterbalanced) prior to moving to the other limb.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-40 years old
* Lower extremity injury-free for at least 3 months
* No previous history of foot or ankle surgery on either limb
* No known history of known foot or ankle fracture on either limb
* No known neurological or vestibular disorders, or other medical conditions affecting balance, including ear infections
* Does not have diabetes mellitus
* No self-reported disability due to lower extremity pathology
* No previous history of ankle sprain on either limb as reported on the Modified Ankle Instability Index questionnaire
* A score lower than 10 on the Identification of Functional Ankle Instability questionnaire

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University and surrounding community
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-08-18 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Balance | 30 second trials
  Force plate derived measures (center of pressure and time to boundary) will be collected.

SECONDARY OUTCOMES:
Cognitive errors | 30 seconds
  The number of cognitive errors during cognitive tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Custer, Ph.D, ATC, Principal Investigator — Towson University
Locations (1):
- Burdick Hall, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 1 year after publication with no end date

REFERENCES:
- [Background] Rahnama L, Salavati M, Akhbari B, Mazaheri M. Attentional demands and postural control in athletes with and without functional ankle instability. J Orthop Sports Phys Ther. 2010 Mar;40(3):180-7. doi: 10.2519/jospt.2010.3188. PMID 20195021